CLINICAL TRIAL: NCT03567642
Title: Phase 1 Study of Combination Osimertinib, Platinum, Etoposide for Patients With Metastatic EGFR Mutant Lung Cancers With Concurrent RB1 and TP53 Alterations
Brief Title: A Study of the Combination of Osimertinib, Platinum and Etoposide for Patients With Metastatic EGFR Mutant Lung Cancers
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-211
Record Dates: First submitted 2018-06-13; First posted 2018-06-26 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Lung Cancer
Keywords: Osimertinib; Platinum; Etoposide; EGFR Mutant; 18-211
MeSH Terms: conditions — Lung Neoplasms | interventions — osimertinib; Platinum; Etoposide

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Osimertinib, Platinum (cisplatin or carboplatin) and Etoposide (Experimental): Initially, 6 patients will be enrolled and will begin treatment with osimertinib 80mg orally daily (3 who will be receiving cisplatin and 3 who will be receiving carboplatin). Cisplatin or carboplatin treatment will be decided by the treating physician prior to study registration. After 9 weeks (+/- 1 week)( 3 cycles) on osimertinib alone, carboplatin or cisplatin and etoposide will be added. Carboplatin is doses at an AUC of 5 or cisplatin at 60mg/m2 will be given on C4D1. Etoposide is dosed at 100mg/m2 given on Days 1-3 of C4. Only patients on osimertinib 80mg orally daily at the start of cycle 4 will be included in the 3+3 dose de-escalation portion of the study. Chemotherapy and osimertinib will be administered concurrently during cycles 4-7, and from cycle 8 onward, osimertinib monotherapy will be continued. Patients will present every 2 cycles post-chemo (Cycles 8, 10, 12, etc.)
  Interventions: Drug: Osimertinib; Drug: Platinum; Drug: Etoposide

INTERVENTIONS:
Drug: Osimertinib — Osimertinib 80mg daily
Drug: Platinum — Cisplatin 60mg/m2 or Cisplatin 45mg/m2 Carboplatin AUC 5 or Carboplatin AUC 4
Drug: Etoposide — Etoposide 100mg/m2 or Etoposide 80mg/m2

SUMMARY:
The purpose of this study is to test the safety of combining Osimertinib with either Cisplatin or Carboplatin (at different dose levels) and Etoposide, to find out what effects, if any, this combination of drugs has on people with EGFR mutant lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Advanced biopsy-proven metastatic non-small cell lung cancer
* Either have not started an EGFR TKI or may have started osimertinib within the last 9 weeks
* Somatic activating mutation in EGFR in pre-treatment tumor biopsy or cfDNA
* Evidence of a concurrent P53 alteration by IHC or NGS on pre-treatment tumor biopsy or cfDNA
* Evidence of a concurrent RB1 alteration by IHC or NGS on pre-treatment tumor biopsy or cfDNA
* Must have a site of disease amenable to repeat biopsy and be willing to undergo a biopsy during treatment
* Measurable (RECIST 1.1) indicator lesion not previously irradiated
* Karnofsky performance status (KPS) ≥ 70%
* Age >18 years old
* Ability to swallow oral medication
* Adequate organ function

  * AST, ALT ≤ 3 x ULN
  * Total bilirubin ≤ 1.5x ULN
  * Creatinine ≤ 1.5x ULN OR calculated creatinine clearance ≥ 60ml/min
  * Absolute neutrophil count (ANC) ≥ 1000 cells/mm^3
  * Hemoglobin≥8.0 g/dL
  * Platelets ≥100,000/mm^3

Exclusion Criteria:

* Pregnant or lactating women
* Started an EGFR TKI other than osimertinib or started osimertinib more than 9 weeks ago
* Any radiotherapy within 1 week of starting treatment on protocol.
* Any major surgery within 1 weeks of starting treatment on protocol.
* Any evidence of active clinically significant interstitial lung disease
* Continue to have unresolved > grade 1 toxicity from any previous treatment
* Have pure small cell histology
* Corrected QT interval using Fridericia's formula (QTcF)>475msec or any clinically significant (as deemed by the investigator) abnormalities in rhythm or conduction or morphology of the resting EKG.
* Patients are to be excluded from cisplatin treatment arm if they meet any of the following criteria:
* Creatinine clearance < 60 ml/min
* Hearing impairment requiring assistive device
* Neuropathy
* The treating provider does not feel as though the patient should receive cisplatin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2018-06-12 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
The MTD (maximum tolerated dose) | 2 years
  Determine the safety and toxicity profile of combination osimertinib, platinum (cisplatin or carboplatin), etoposide for patients with metastatic EGFR mutant lung cancers with concurrent RB1 and TP53 alterations.

CONTACTS AND LOCATIONS:
Overall Officials: Helena Yu, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Cancer Center, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm